CLINICAL TRIAL: NCT00497211
Title: Intracoronary Infusion of BM-Derived Mononuclear Cells in Patients With Large Acute Myocardial Infarction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Antwerp (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC 3/39/123
Record Dates: First submitted 2007-07-04; First posted 2007-07-06 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Myocardial Infarction
Keywords: First large acute myocardial infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Intracoronary mononuclear cell infusion

SUMMARY:
Large acute myocardial infarctions are the most frequent cause of subsequent systolic heart failure. Some evidence exists on the improvement after intracoronary administration of bone marrow cells in patients with a recente acute myocardial infarction. Although subgroup analyses suggest that patients with the largest myocardial infarctions have the largest increase in ejection fraction after intracoronary bone marrow administration, there is no published trial including only large myocardial infarctions. Therefor we sought to confirm the subgroup analyses by conducting a trial in only large first acute myocardial infarction patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 and <80 years old
* Acute myocardial infarction >2 and <96 hours from start to reperfusion
* Cumulative ST-segment elevation >6 mm on 12 lead ECG
* No functional myocardial impairment outside the myocardial infarction region
* Succesful PCI of infarct related coronary artery
* Left ventricular ejection fraction <50% on ventriculography, echo or MRI
* Accepted anticonceptive use during the study for women of childbearing potential
* Written and signed informed consent

Exclusion Criteria:

* CPR > 10 minuts or persistent cardiogenic shock
* complete left bundle branch block without concordant ST-segment elevation
* Need foor cardiac surgery (valvular, coronary or other)
* Trombocytopenia, coagulation disorders or hematological disease
* History or active malignancy
* Life expectancy (apart from acute myocardial infarction) <5 years
* Dialysis or severe kidney insufficiency (creatinin clearance <30ml/')
* Severe liver insufficiency
* Severe respiratory disease
* Systemic inflammatory pathology (acute or chronic, apart from inflammation associated with myocardial infarction)
* Symptomatic cerebral or periferal vascular disease
* Prior myocardial infarction or prior myocardial dysfunction
* Prior CABG or heart valve surgery
* Pregnancy, pregnancy wish or lactation <1 month
* Psychiatrical illness
* Physical or psychological inability to adhere to the protocol
* Participation in other not yet completed study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Steven E Haine, MD, Principal Investigator — UZ Antwerpen; Chris Vrints, MD, PhD, Study Director — UZ Antwerpen
Locations (1):
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium